CLINICAL TRIAL: NCT04939987
Title: Opioid-Free Pain Control Regiment Following Robotic Radical Prostatectomy: A Randomized Controlled Trial
Brief Title: Opioid-Free Pain Control Regiment Following Robotic Radical Prostatectomy
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI left institution and study was not transferred to new PI
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00074034
Record Dates: First submitted 2021-06-01; First posted 2021-06-25 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-05

CONDITIONS: Radical Prostatectomies
Keywords: opioids; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Analgesics, Opioid; Gabapentin; oxycodone-acetaminophen; Ketorolac; Acetaminophen; Ketorolac Tromethamine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Control Cohort (Active Comparator): One treatment selected:
  Tramadol (50mg) Hydrocodone-Acetaminophen (2.5mg/325mg) Oxycodone-Acetaminophen (2.5mg/325mg)
  Interventions: Drug: Tramadol; Drug: Hydrocodone-Acetaminophen; Drug: Oxycodone-Acetaminophen
- Experimental Cohort (Experimental): Multimodal Approach:
  Gabapentin (100mg TID) Ketorolac (15mg q6) Acetaminophen (1mg IV q6) Ketamine (1.5mg/kg) Ketorolac tromethamine (15mg or 30mg Q4)
  Interventions: Drug: Gabapentin; Drug: Ketorolac; Drug: Acetaminophen; Drug: Ketorolac tromethamine; Drug: Ketamine

INTERVENTIONS:
Drug: Tramadol — Opioid Control Cohort (One treatment selected)
  Other Names: Opioid
  Arms: Opioid Control Cohort
Drug: Gabapentin — Experimental Cohort (Multimodal Approach)
  Arms: Experimental Cohort
Drug: Hydrocodone-Acetaminophen — Opioid Control Cohort (One treatment selected)
  Other Names: Opioid
  Arms: Opioid Control Cohort
Drug: Oxycodone-Acetaminophen — Opioid Control Cohort (One treatment selected)
  Other Names: Opioid
  Arms: Opioid Control Cohort
Drug: Ketorolac — Experimental Cohort (Multimodal Approach)
  Arms: Experimental Cohort
Drug: Acetaminophen — Experimental Cohort (Multimodal Approach)
  Arms: Experimental Cohort
Drug: Ketorolac tromethamine — Experimental Cohort (Multimodal Approach)
  Arms: Experimental Cohort
Drug: Ketamine — Experimental Cohort (Multimodal Approach)
  Arms: Experimental Cohort

SUMMARY:
This study will address the gaps in research of non-opioid postoperative pain management for prostatectomies.

DETAILED DESCRIPTION:
This study will conduct a randomized control double-blind clinical trial to evaluate an opioid versus a non-opioid pathway of gabapentin, ketorolac, and acetaminophen in treating postoperative pain following robot-assisted radical prostatectomy (RARP).

ELIGIBILITY:
Inclusion Criteria:

* All men ages 40-75 undergoing bilateral robot assisted radical prostatectomy (RARP) with bilateral lymph node dissection with low-intermediate to high-risk localized prostate cancer

Exclusion Criteria:

* Allergies to any medication involved in the study
* T4 prostate cancer
* incarcerated persons
* chronic narcotic dependence
* any current prescription for narcotics
* any surgery in the past 6 months

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Pain Score | 1 hour before surgery
  Pain scores will be collected using the Visual Analogue Pain Score and measured on a scale of 0-10, with 0 being no pain 10 being the worst pain imaginable
Visual Analogue Pain Score | Baseline
  Pain scores will be collected using the Visual Analogue Pain Score and measured on a scale of 0-10, with 0 being no pain 10 being the worst pain imaginable
Visual Analogue Pain Score | Day 1
  Pain scores will be collected using the Visual Analogue Pain Score and measured on a scale of 0-10, with 0 being no pain 10 being the worst pain imaginable
Visual Analogue Pain Score | Day 3
  Pain scores will be collected using the Visual Analogue Pain Score and measured on a scale of 0-10, with 0 being no pain 10 being the worst pain imaginable
Visual Analogue Pain Score | Day 7
  Pain scores will be collected using the Visual Analogue Pain Score and measured on a scale of 0-10, with 0 being no pain 10 being the worst pain imaginable
Amount of medication used | 1 hour before surgery
  measure opioid utilization by surveying patients on their usage while collecting their pain scores - Opioid oral morphine milligram equivalents (OMEQ) will be measured
Amount of medication used | Baseline
  measure opioid utilization by surveying patients on their usage while collecting their pain scores - Opioid oral morphine milligram equivalents (OMEQ) will be measured
Amount of medication used | Day 1
  measure opioid utilization by surveying patients on their usage while collecting their pain scores - Opioid oral morphine milligram equivalents (OMEQ) will be measured
Amount of medication used | Time of Discharge postoperative up to Day 3
  measure opioid utilization by surveying patients on their usage while collecting their pain scores - Opioid oral morphine milligram equivalents (OMEQ) will be measured
Opioid-Related Symptom Distress Scale (ORSDS) | 1 hour before surgery
  4-point scale that evaluates 12 symptoms in 3 symptom categories including frequency, severity, and bothersomeness. The ORSDS may be used to calculate a symptom-specific score, which is the average of the 3 symptom distress dimensions and range from 0 to 4. The composite ORSDS score is the mean of all 12 symptom-specific scores. Composite ORSDS scores range from 0 to 4.
Opioid-Related Symptom Distress Scale (ORSDS) | Baseline
  4-point scale that evaluates 12 symptoms in 3 symptom categories including frequency, severity, and bothersomeness. The ORSDS may be used to calculate a symptom-specific score, which is the average of the 3 symptom distress dimensions and range from 0 to 4. The composite ORSDS score is the mean of all 12 symptom-specific scores. Composite ORSDS scores range from 0 to 4.
Opioid-Related Symptom Distress Scale (ORSDS) | Day 1
  4-point scale that evaluates 12 symptoms in 3 symptom categories including frequency, severity, and bothersomeness. The ORSDS may be used to calculate a symptom-specific score, which is the average of the 3 symptom distress dimensions and range from 0 to 4. The composite ORSDS score is the mean of all 12 symptom-specific scores. Composite ORSDS scores range from 0 to 4.
Opioid-Related Symptom Distress Scale (ORSDS) | Day 3
  4-point scale that evaluates 12 symptoms in 3 symptom categories including frequency, severity, and bothersomeness. The ORSDS may be used to calculate a symptom-specific score, which is the average of the 3 symptom distress dimensions and range from 0 to 4. The composite ORSDS score is the mean of all 12 symptom-specific scores. Composite ORSDS scores range from 0 to 4.
Opioid-Related Symptom Distress Scale (ORSDS) | Day 7
  4-point scale that evaluates 12 symptoms in 3 symptom categories including frequency, severity, and bothersomeness. The ORSDS may be used to calculate a symptom-specific score, which is the average of the 3 symptom distress dimensions and range from 0 to 4. The composite ORSDS score is the mean of all 12 symptom-specific scores. Composite ORSDS scores range from 0 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Ram Pathak, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No